CLINICAL TRIAL: NCT04117412
Title: The Oxidative Stress, Inflammatory Markers, and Metabolomics Response to Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Oxidative Stress, Inflammatory Markers, and Metabolomics Response to Exercise in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Research Assistant, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GO 18/1121-05
Record Dates: First submitted 2019-09-05; First posted 2019-10-07 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Same participants will undergo two different exercise protocols after maximal exercise test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with COPD (Other): Patients with COPD will undergo two different one bout of exercise training after maximal exercise test.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Same participants will undergo different one bout of exercise protocols

SUMMARY:
The effect of different physical exercise protocols on inflammatory markers, antioxidant balance, and metabolomics has not been fully elucidated. Therefore, the purpose of this study is to investigate the responses of oxidative stress, inflammatory markers, and metabolomics to exercise.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD), one of the major causes of morbidity and mortality, is a preventable and curable disease characterized by irreversible airflow limitation. The progressive lung involvement, systemic inflammation, respiratory and peripheral muscle dysfunction, loss of muscle mass, and the dysfunction of the remaining muscles occur in COPD. Muscle dysfunction, which is defined as loss of strength or loss of endurance characteristics in muscles, is a comorbidity associated with poor outcomes such as frequent hospitalization and decreased survival, as well as adversely affecting exercise capacity and quality of life. Exercise increases mitochondrial activity and requires antioxidant defense to achieve cellular redox regulation. The effect of different physical exercise protocols on inflammatory markers, antioxidant balance, and metabolomics has not been fully elucidated. Oxidative stress, inflammatory markers, and metabolic responses to different acute exercise modalities in COPD patients need to be examined and clarified. Therefore, the purpose of this study is to investigate the responses of oxidative stress, inflammatory markers, and metabolomics to exercise. Detection of biomolecules that change with acute exercise may also contribute to the identification of exercise-related pathways.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (clinically stable)
* Being 40-80 years of age
* Able and willing to complete the informed consent process.

Exclusion Criteria:

* To have severe neuromuscular, musculoskeletal and rheumatic problems
* Unable to cooperate

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Response of total work values to maximal exercise test, high intensity interval and continuous exercise | Change from baseline to after maximal exercise test, high intensity interval, and continuous exercise, up to 3 weeks.
  Peak work rates will be determined using cycle ergometer. Maximal exercise test will be performed on the first day, high intensity interval and continuous exercise will be performed with one week intervals.
The inflammatory markers response to maximal exercise test, high intensity interval and continuous exercise | Change from baseline to after maximal exercise test, high intensity interval, and continuous exercise, up to 3 weeks.
  Blood samples will be collected before and after exercise and analyzed for the responses of IL-1, IL-6, TNF-α, sTNFr1. Maximal exercise test will be performed on the first day, high intensity interval and continuous exercise will be performed with one week intervals.
The oxidative response to maximal exercise test, high intensity interval and continuous exercise | Change from baseline to after maximal exercise test, high intensity interval, and continuous exercise, up to 3 weeks.
  Blood samples will be collected before and after exercise and analyzed for the responses of glutathione peroxidase, catalase, superoxide dismutase, glutathione, and total antioxidant status. Maximal exercise test will be performed on the first day, high intensity interval and continuous exercise will be performed with one week intervals.
The metabolomics response (valine-leucine-isoleucine, alanine) to maximal exercise test, high intensity interval, and continuous exercise. | Change from baseline to after maximal exercise test, high intensity interval, and continuous exercise, up to 3 weeks.
  Blood samples will be collected before and after exercise and analyzed for identification of metabolomics which change with exercise. Maximal exercise test will be performed on the first day, high intensity interval and continuous exercise will be performed with one week intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, Study Director — Hacettepe University; Aslihan Cakmak, MSc, Principal Investigator — Hacettepe University; Emirhan Nemutlu, PhD, Principal Investigator — Hacettepe University; Samiye Yabanoglu-Ciftci, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Cakmak A, Nemutlu E, Yabanoglu-Ciftci S, Baysal I, Kocaaga E, Coplu L, Inal-Ince D. Metabolomic, oxidative, and inflammatory responses to acute exercise in chronic obstructive pulmonary disease. Heart Lung. 2023 May-Jun;59:52-60. doi: 10.1016/j.hrtlng.2023.01.011. Epub 2023 Jan 30. PMID 36724589